CLINICAL TRIAL: NCT00237939
Title: A Prospective, Multicenter, Open-Label Study of Aripiprazole in the Management of Patients With Schizophrenia in General Psychiatric Practices (Broad Effectiveness Trial With Aripiprazole- BETA)
Brief Title: A Study of Aripiprazole in the Management of Patients With Schizophrenia in the General Psychiatric Practices
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka America Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CN138-100
Record Dates: First submitted 2005-10-11; First posted 2005-10-13 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2007-10

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole

SUMMARY:
The purpose of this clinical research study is to evaluate if Aripiprazole will prove to be effective, safe and well tolerated in the treatment of patients with schizophrenia who are treated in a general psychiatric setting.

ELIGIBILITY:
Inclusion Criteria:

* Clinical DSM-IV diagnosis of schizophrenia
* Patients being managed as outpatients, for whom an alteration in medication is clinically reasonable or initiation of antipsychotics is required

Exclusion Criteria:

* Risk of committing suicide, diagnosis of schizoaffective disorder, bipolar disorder, depression with psychotic syptoms, or organic brain syndromes
* Prisoners or subjects compulsory detained

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200
Dates: Start 2002-09; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression-Improvement at endpoint

SECONDARY OUTCOMES:
Patients' and caregivers' medication preference

CONTACTS AND LOCATIONS:
Overall Officials: Hervé Allain, MD, Principal Investigator — Faculté de Médecine de Rennes I, laboratoire de pharmacologie
Locations (20):
- Belgium (9):
  - Local Institution, Antwerp
  - Local Institution, Brussels
  - Local Institution, Diest
  - Local Institution, Kortenberg
  - Local Institution, Liège
  - Local Institution, Sint-Michiels
  - Local Institution, Sint-Niklaas
  - Local Institution, Sint-Truiden
  - Local Institution, Tournai
- Local Institution, Rennes, France
- Netherlands (3):
  - Local Institution, Amersfoort
  - Local Institution, Raalte
  - Local Institution, Rotterdam
- Portugal (4):
  - Local Institution, Barcelos
  - Local Institution, Ceira
  - Local Institution, Coimbra
  - Local Institution, Lisbon
- Spain (3):
  - Local Institution, Barcelona
  - Local Institution, Salamanca
  - Local Institution, Seville